CLINICAL TRIAL: NCT00820937
Title: Interest of the Combination of the DaTSCAN Scintigraphy and MRI Scan in the Differential Diagnosis of Lewy Body Dementia From Alzheimer Disease in Patients With Hallucinations
Brief Title: Diagnostic of Lewy Body Dementia by Combining Scintigraphy (SPECT) Using a Specific Transporter and Magnetic Resonance Imaging (MRI)
Acronym: DatScan
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Limoges (Other)
Responsible Party: Marie SENGELEN, CHU Limoges
Allocation: Not Applicable | Model: Single Group | Purpose: Diagnostic
Other Study IDs: I04014
Record Dates: First submitted 2008-12-27; First posted 2009-01-12 (Estimated); Last update posted 2025-07-30 (Actual); Status verified 2009-08

CONDITIONS: Lewy Body Dementia
MeSH Terms: conditions — Lewy Body Disease | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Single photon emission computed tomography and Magnetic Resonance Imaging

SUMMARY:
The aim of this study is to improve the diagnostic of Lewy body dementia by combining the scintigraphy (SPECT) usig a spécific transporter and magnetic resonance imaging (MRI).

DETAILED DESCRIPTION:
Lewy body dementia is the second leading cause of dementia in France after degenerative Alzheimer's disease.

However its dignosis is difficult. Its comes in large part from the similarity of symptoms with another close dementia syndrome : the Alzheimer disease . Therfore, its is very important to have a mean to distinguish between the two dementias.

One highlight of the Lewy body dementia process being dopaminergic degeneration, the use of specific radioactive tracers is thought to be the way. The radiotracer that has the greatest advantage for these explorations is currently the DaTSCAN because it binds specifically on the dopamine transporter and can be used in Single photon emission computed tomography (SPECT).

The aim of this study is to improve the performance of imaging in the diagnosis of dementia by combining scintigraphy (SPECT) and magnetic resonance imaging (MRI) in the exploration of the striatal region . The development of this method applied to a population of subjects, with hallucinations and cognitive disorders, should demonstrate the value and complementarity of metabolic images (SPECT) and morphological (MRI) within the differential diagnosis of Lewy body dementia and the Alzheimer disease .

From a methodological point of view, the patient will be included in hospital and will have a clinical diagnosis defined according to the criteria of dementia NINCDS-ADRDA for the Alzheimer disease and Mc-Keith criteria for Lewy body dementia. Their MMSE will be over 18 and they have in common recurrent visual hallucinations.

After the inclusion, two steps must be distinguished, a neuropsychological evaluation stage and an scitigraphy exploration . Before the SPECT , all patients should have an MRI.

ELIGIBILITY:
Inclusion Criteria:

* Patients with alzheimer disease following NINCDS-ADRDA scale or Lewy body dementia following Mc Keith scale.
* Aged between 65 et 90 years
* Patients with visual hallucination
* Patients with helping people
* Patients with MMSE (Mini Mental State Examination) equal or more than 18.
* Signed consent

Exclusion Criteria:

* Hospitalized patients without their consent
* Patients who have not passed the neuropsychological tests
* Patients with a MMSE less than 18
* Patients without helping
* Patients with no visual hallucinations
* Patients with severe somatic pathology.
* Pregnancy
* Allergy to iodine

Ages: 65 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 20 (Actual)
Dates: Start 2006-03; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
SPECT and MRI differential imaging | Visit 1

SECONDARY OUTCOMES:
Neuropsychological analysis | Visit 1

CONTACTS AND LOCATIONS:
Locations (3):
- France (3):
  - Département de Gérontologie - Chu Limoges, Limoges
  - Pôle de psychiatrie du sujet âgé - CH Esquirol, Limoges
  - Service de Neurologie - CHU de Limoges, Limoges

REFERENCES:
- [Result] Comparison of DAT-scan evaluation for the aetiological diagnosis of hallucinations in the elderly P. Thomas a,∗,d, A. Prado-Jeana,b, J.-P. Clément a,d, P. Couratier a,b, J. Monteil c NPG Neurologie - Psychiatrie - Gériatrie Volume 13, Issue 75, June 2013, Pages 145-151